CLINICAL TRIAL: NCT02055105
Title: Modulation of Molecular Fingerprinting in Pediatric Sepsis
Status: Recruiting | Type: Observational
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PHNX-biosep-12159
Record Dates: First submitted 2014-01-27; First posted 2014-02-04 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: Pediatric Sepsis
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Biospecimen Retention: Samples With DNA — Blood samples, urine samples and buccal swabs will be obtained from these patients at 5 time points to analyze biomarkers. Study participants will receive standard of care with antimicrobials and any additional appropriate cardiovascular or respiratory support per the clinical team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 10 Patients with sepsis or septic shock: Previously healthy, non-immunocompromised patients, between the ages of 1 and 18, who are being admitted to the PCH PICU for sepsis or septic shock, will be enrolled. Blood samples, urine samples and buccal swabs will be obtained from these patients at 5 time points to analyze biomarkers. Study participants will receive standard of care with antimicrobials and any additional appropriate cardiovascular or respiratory support per the clinical team. The samples will collected and stored at -80 until analysis can be performed. In addition to, during the course of the hospitalization, the enrolled patient will have data collected to calculate severity scores, including PRISM scores and TISS-28 scores. All patient information will be de-identified. A standard procedure manual will be developed detailing the methods for data collection and entry.
  Interventions: Procedure: miRNA in Sepsis
- 50 Healthy Patients: Healthy non-immunocompromised patients between 1-18 years old

INTERVENTIONS:
Procedure: miRNA in Sepsis — miRNA in Sepsis
  Groups: 10 Patients with sepsis or septic shock

SUMMARY:
The goal of this study is to demonstrate the sensitivity and specificity of detecting circulating micro RNA (miRNA) biomarkers in pediatric septic patients. It will also follow expression and modulation of levels in response to therapy in comparison to current biomarkers.

DETAILED DESCRIPTION:
This study will aid in the evaluation of determining the accuracy of these miRNAs in pediatric patients and help in establishing pilot data for additional studies in the future. The testing will include blood samples, urine samples and buccal swabs from patients who meet eligibility at 5 time points to analyze biomarkers. Study participants will receive standard of care with antimicrobials and any additional appropriate cardiovascular or respiratory support per the clinical team. The samples will collected and stored at -80 until analysis can be performed. In addition to, during the course of the hospitalization, the enrolled patient will have data collected to calculate severity scores, including updated Pediatric Risk of Mortality (PRISM III) scores and simplified Therapeutic Intervention Scoring System(TISS-28) scores. All patient information will be de-identified. A standard procedure manual will be developed detailing the methods for data collection and entry. Data will be recorded in a de-identified manner on a Microsoft Excel database on a secure institutional server by the institutional staff. Data will then be analyzed to determine correlation of biomarkers to morbidity and mortality for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 through 18 years
* Patients admitted to the PICU with concerns for sepsis or those developing sepsis during their admission to the hospital.
* Patients must be enrolled int he study from arrival time tot he ED up to 24 hours from the time of initiation of antibiotic therapy for treatment of sepsis or septic shock.
* Signed informed consent.

Exclusion Criteria:

* Patients <1 year of age and greater than 18 years of age.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children ages 1-18 who are Immune-competent (no previous chronic medical conditions) patients being admitted to the PICU at PCH with concerns for sepsis or those developing sepsis during their admission to the hospital who require care in the PICU.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Risk of Mortality | Duration of hospital stay, an expected average of 3 weeks
  Will compare PRISM 3 scores from baseline to hospital discharge.

SECONDARY OUTCOMES:
Organ Failure | Duration of hospital stay, an expected average of 3 weeks
  Will compare sequential organ failure assessment (SOFA) scores throughout hospitalization.
Organ Dysfunction | Duration of hospital stay, an expected average of 3 weeks
  Will compare pediatric multiple organ dysfunction scores (PMODS) throughout hospitalization
Patient acuity | Duration of hospital stay, an expected average of 3 weeks
  Will assess TISS-28 scores throughout hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Willyerd, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Principal investigator is undecided if he plans on having a DTA or MTA.